CLINICAL TRIAL: NCT00949468
Title: Epidemiologic Characteristics, Predisposing Factors and Microbiological Profile of Infectious Corneal Ulcers in Two Referral Centers in a Countryside City of Brazil
Brief Title: Microbiological Keratitis in a Countryside City of Brazil
Status: Completed | Type: Observational
Sponsor: Sao Jose do Rio Preto Medical School (Other)
Collaborators: Conselho Nacional de Desenvolvimento Científico e Tecnológico (Other Government)
Responsible Party: Thiago Lopes Genaro, Sao Jose do Rio Preto University
Other Study IDs: Opht2009
Record Dates: First submitted 2009-07-29; First posted 2009-07-30 (Estimated); Last update posted 2009-07-30 (Estimated); Status verified 2009-07

CONDITIONS: Keratitis
Keywords: Keratitis
MeSH Terms: conditions — Keratitis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Corneal scrapes
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Keratitis group: 37 patients with keratitis
- Control Study Group: 37 control volunteers

SUMMARY:
The purpose of this study is to identify the predisposing factors, epidemiological features and clinical and microbiological diagnosis of infectious keratitis in two public referral centers of ophthalmology in a countryside city of Brazil.

ELIGIBILITY:
Inclusion Criteria:

* All patients admitted with clinical suspicious of keratitis from June 2008 to June 2009 (Keratitis group)
* 37 volunteers without any ophthalmologic claim, recruited in the two ophthalmology centers listed (Control study group)

Exclusion Criteria:

* In the Control Study Group, no infectious ocular disease was accepted

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: 37 patients admitted in two referral ophthalmology centers in a countryside city of Brazil. 37 volunteers were used as a control group.
Sampling Method: Non-Probability Sample
Enrollment: 74 (Actual)
Dates: Start 2008-06; Primary Completion 2009-06 (Actual); Study Completion 2009-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Thiago Lo Genaro, Academic, Principal Investigator — Sao Jose do Rio Preto Medical School
Locations (1):
- Sao Jose do Rio Preto University, São José do Rio Preto, São Paulo, Brazil